CLINICAL TRIAL: NCT06606535
Title: ENDO-BRAIN: Effects of Endocrine Adjuvant Therapy with Aromatase Inhibitors on the Cognitive Function of Breast Cancer Patients
Acronym: ENDO-BRAIN
Status: Recruiting | Type: Observational
Sponsor: Ospedale Policlinico San Martino (Other)
Collaborators: University of Genova (Other)
Responsible Party: Principal Investigator, Claudia Massarotti, Principal Investigator, Ospedale Policlinico San Martino
Other Study IDs: ENDO-BRAIN; DB id 13624 (Other: regional IRB (CERLiguria))
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Side Effects of Cancer Therapy; Hypoestrogenism
Keywords: breast cancer; cognitive side effects; hypoestrogenism; ovarian function suppression; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Breast cancer patients undergoing endocrine adjuvant therapy with Aromatase Inhibitors (+ GnRH analogues if they are premenopausal)
  Interventions: Diagnostic Test: validated questionnaires; Diagnostic Test: functional MRI; Diagnostic Test: Optical Coherent Tomography Angiography
- Controls: Healthy age-matched women who are not using hormonal contraception or hormonal replacement therapy at the time of the study.
  Interventions: Diagnostic Test: validated questionnaires; Diagnostic Test: functional MRI; Diagnostic Test: Optical Coherent Tomography Angiography

INTERVENTIONS:
Diagnostic Test: validated questionnaires — Validated questionnaires for climacteric symptoms
Diagnostic Test: functional MRI — functional MRI
Diagnostic Test: Optical Coherent Tomography Angiography — OCT angiography, macular and peripapillary scans
  Other Names: OCT angiography

SUMMARY:
The principal aim of this prospective observational study is to investigate the cognitive function of breast cancer patients that use AI, comparing it with age-matched healthy controls, utilizing cognitive assessments and functional magnetic resonance imaging (fMRI). Additionally, the project seeks to establish correlations between cognitive function and other estrogen deprivation symptoms, including vasomotor symptoms, and to evaluate a possible correlation with endothelial damage studied through Angio Optical Coherent Tomography (angio OCT).

Patients will be recruited during follow up visits at the iatrogenic menopause outpatient clinic. After informed consent, the will be asked for detailed demographic data, medical, oncological and gynecological history. Hypoestrogenism symptoms will be collected through validated questionnaires. The cognitive assessment will be performed on the same day, by trained staff. The fMRI and angioOCT will be booked and performed depending on patient and clinic availability.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients undergoing endocrine adjuvant therapy with AI, with or without GnRH agonists, depending on menopause status at diagnosis (cases only)
* At least 18 years old
* Good comprehension of oral and written Italian language

Exclusion Criteria:

* incomplete ovarian suppression (cases)
* previous neoplastic diseases other than the presently treated breast cancer for cases
* known neurological or psychiatric disorders
* use of hormonal contraception or hormonal replacement therapy (controls)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a monocentric study, taking place in an university hospital, which is a referral point for both oncology and neurology.
  Cases are recruited from the iatrogenic menopause outpatient clinic. This is a dedicated outpatient clinic for the gynecological follow up of cancer survivors, including breast cancer patients undergoing adjuvant endocrine therapy. It is part of the oncofertility pathway of the institution, it is run by doctors with specific expertise in reproductive endocrinology, fertility and menopause. The clinic is accessed by all patients, not only the symptomatic ones, for yearly follow ups. Healthy controls are recruited from the gynecological, neurological or ophthalmological outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
cognitive assessment | Once, at enrollment.
  The principal aim of this project is to investigate the cognitive function of breast cancer patients that use Aromatase Inhibitors, comparing it with age-matched healthy controls, utilizing cognitive assessment and fMRI.
  * neuropsychological battery composed of the i) prose recall test, ii) trail making test A and B, iii) digit span backward and forward and iv) the symbol digit modalities test
  * 3T MRI (Siemens Prisma): 3D sagittal T2-FLAIR; 3D MP2RAGE; T2* gradient echo-planar imaging under resting condition; twice-refocused spin echo echo-planar imaging sequence for multi-shell diffusion-weighted images

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Policlinico San Martino, Genova, GE, Italy

REFERENCES:
- [Background] Menning S, de Ruiter MB, Veltman DJ, Boogerd W, Oldenburg HS, Reneman L, Schagen SB. Changes in brain activation in breast cancer patients depend on cognitive domain and treatment type. PLoS One. 2017 Mar 7;12(3):e0171724. doi: 10.1371/journal.pone.0171724. eCollection 2017. PMID 28267750
- [Background] Chen X, He X, Tao L, Li J, Wu J, Zhu C, Yu F, Zhang L, Zhang J, Qiu B, Yu Y, Wang K. The Working Memory and Dorsolateral Prefrontal-Hippocampal Functional Connectivity Changes in Long-Term Survival Breast Cancer Patients Treated with Tamoxifen. Int J Neuropsychopharmacol. 2017 May 1;20(5):374-382. doi: 10.1093/ijnp/pyx008. PMID 28177081